CLINICAL TRIAL: NCT06741124
Title: Comparison of Channel Esophagogastrostomy and Double Tract Reconstruction After Laparoscopic-assist Proximal Gastrectomy: a Propensity Score-Matched Analysis
Status: Completed | Type: Observational
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NorthernJiangsuCEDTR; CEDTR (Other: CEDTR)
Record Dates: First submitted 2024-12-16; First posted 2024-12-18 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2020-09

CONDITIONS: Gastric (Stomach) Cancer
Keywords: Proximal Gastrectomy; Channel Esophagogastrostomy; Double Tract Reconstruction
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Channel Esophagogastrostomy (CE): Patients who underwent Channel Esophagogastrostomy reconstruction
  Interventions: Procedure: Channel Esophagogastrostomy
- Double Tract Reconstruction (DTR): Patients who underwent DTR reconstruction during LAPG
  Interventions: Procedure: Double Tract Reconstruction

INTERVENTIONS:
Procedure: Channel Esophagogastrostomy — Channel Esophagogastrostomy
  Groups: Channel Esophagogastrostomy (CE)
Procedure: Double Tract Reconstruction — Double Tract Reconstruction
  Groups: Double Tract Reconstruction (DTR)

SUMMARY:
This retrospective cohort study enrolled adult patients who underwent LAPG between September 2020 and September 2023 at Northern Jiangsu People's Hospital. Patients were categorized into the CE group (CE anastomosis) and the DTR group (DTR anastomosis) based on the digestive tract reconstruction method after LAPG. Variables such as sex and BMI may influence the technical difficulty and clinical outcomes of LAPG. To minimize bias, propensity score (PS) matching was performed at a 1:2 ratio between the CE group and the DTR group.

DETAILED DESCRIPTION:
This retrospective cohort study enrolled adult patients who underwent LAPG between September 2020 and September 2023 at Northern Jiangsu People's Hospital. This study was approved by the Medical Ethics Committee of Northern Jiangsu People's Hospital, and the requirement for written informed consent was waived due to the retrospective study design. This study adhered to the STROCSS 2021 guidelines and was conducted in accordance with the Declaration of Helsinki. The inclusion criteria were as follows: (1) Patients with a malignant tumor in the upper one-third of the stomach, diagnosed through endoscopy and pathology, with no distant metastases confirmed by multislice spiral computed tomography, and who underwent elective LAPG; (2) Patients who underwent CE reconstruction or DTR during LAPG; and (3) Patients available for postoperative follow-up. The exclusion criteria were as follows: (1) Patients who had received neoadjuvant radiotherapy or chemotherapy prior to surgery; (2) Emergency surgery patients; (3) Patients with concurrent malignancies; (4) Lost to follow-up patients. All surgeries were conducted by the same surgical team. Before the procedure, patients were comprehensively informed about their condition and the surgical approach. After a detailed explanation of the two digestive tract reconstruction methods, the choice between CE or DTR anastomosis was made in accordance with each patient's preference. Patients were categorized into the CE group (CE anastomosis) and the DTR group (DTR anastomosis) based on the digestive tract reconstruction method after LAPG. Variables such as sex and BMI may influence the technical difficulty and clinical outcomes of LAPG. To minimize bias, propensity score (PS) matching was performed at a 1:2 ratio between the CE group and the DTR group, based on age, sex, preoperative BMI, American Society of Anesthesiologists (ASA) score, and history of abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

(1) Patients with a malignant tumor in the upper one-third of the stomach, diagnosed through endoscopy and pathology, with no distant metastases confirmed by multislice spiral computed tomography, and who underwent elective LAPG; (2) Patients who underwent CE reconstruction or DTR during LAPG; and (3) Patients available for postoperative follow-up.

Exclusion Criteria:

(1) Patients who had received neoadjuvant radiotherapy or chemotherapy prior to surgery; (2) Emergency surgery patients; (3) Patients with concurrent malignancies; (4) Lost to follow-up patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients who underwent LAPG between September 2020 and September 2023 at Northern Jiangsu People's Hospital. Patients who underwent CE reconstruction or DTR during LAPG;
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Endoscopic reflux esophagitis | Postoperative one year
  Los Angeles classification

SECONDARY OUTCOMES:
PGSAS-45 questionnaires | Postoperative one year
  Postgastrectomy syndrome assessment scale (PGSAS-45) developed by the Japanese Post-Gastrectomy Symptom Assessment Study Group, is used to objectively evaluate postoperative symptom, quality of life of patients after gastrectomy. It reflects symptoms in seven areas: gastroesophageal reflux, abdominal pain, meal-related distress, dyspepsia, diarrhea, constipation, and dumping syndrome.

OTHER OUTCOMES:
Nutritions status | Postoperative one month, Postoperative three month, Postoperative nine month, Postoperative twelve month,
  alb, hb,

CONTACTS AND LOCATIONS:
Locations (1):
- Northern Jiangsu People's Hospital, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided
Data that support the findings of this study are available from the corresponding author upon reasonable request.

REFERENCES:
- [Background] Liu K, Yang K, Zhang W, Chen X, Chen X, Zhang B, Chen Z, Chen J, Zhao Y, Zhou Z, Chen L, Hu J. Changes of Esophagogastric Junctional Adenocarcinoma and Gastroesophageal Reflux Disease Among Surgical Patients During 1988-2012: A Single-institution, High-volume Experience in China. Ann Surg. 2016 Jan;263(1):88-95. doi: 10.1097/SLA.0000000000001148. PMID 25647058
- [Derived] Zhou J, Li R, Cheng Y, Zhao S, Wang J, Fu Y, Tian Z, Wang L, Wang W, Ren J, Wang D. Comparison of channel esophagogastrostomy and double tract reconstruction after laparoscopic-assisted proximal gastrectomy: a propensity score-matched analysis. Surg Endosc. 2025 Sep;39(9):5722-5732. doi: 10.1007/s00464-025-11978-w. Epub 2025 Jul 17. PMID 40676300